CLINICAL TRIAL: NCT00496054
Title: Evaluation of Safety,Tolerability and Immunogenicity of Vaccination With Rotateq (V260) in Healthy Infants in India
Brief Title: Safety,Tolerability and Immunogenicity of Vaccination With Rotateq in Healthy Infants in India (V260-021)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V260-021; 2007_020
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2010-03-11 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Gastroenteritis; Rotavirus
MeSH Terms: conditions — Gastroenteritis | interventions — Rotavirus Vaccines

ARMS (1):
- RotaTeq™ Vaccine (V260) (Experimental): Evaluation of Safety, Tolerability and Immunogenicity of Vaccination with RotaTeq™ in Healthy Infants in India.
  Interventions: Biological: Rotavirus Vaccine, Live, Oral, Pentavalent

INTERVENTIONS:
Biological: Rotavirus Vaccine, Live, Oral, Pentavalent — Pentavalent vaccine 9G1, G2, G3, G4 & P1) given 3 times. Dose 1 will be administered at study entry; Dose 2 will be administered 4 to 10 weeks (28 to 70 days) after Dose 1; and Dose 3 will be administered 4 to 10 weeks (28 to 70 days) after Dose 2.
  Other Names: RotaTeq™ Vaccine; V260

SUMMARY:
To observe the safety, tolerability and immunogenicity of the administration of 3 doses of rotateq in healthy Indian infants between 6 weeks through exactly 12 weeks of age at entry.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 weeks through exactly 12 weeks
* Healthy infants

Exclusion Criteria:

* Clinical evidence of active gastrointestinal illness
* Fever, with a rectal temperature of greater than and equal to thirty eight degree celsius at the time of immunization
* History of congenital abdominal disorders, intussusception, or abdominal surgery
* History of known prior rotavirus disease
* Known or suspected impairment of immunological function
* Prior administration of any rotavirus vaccine
* Known hypersensitivity to any component of the rotavirus vaccine, e.g. trypsin

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Lokeshwar MR, Bhave S, Gupta A, Goyal VK, Walia A. Immunogenicity and safety of the pentavalent human-bovine (WC3) reassortant rotavirus vaccine (PRV) in Indian infants. Hum Vaccin Immunother. 2013 Jan;9(1):172-6. doi: 10.4161/hv.22341. PMID 23442588

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III
  First Patient In (FPI): 09-May-2008
  Last Patient Out (LPO): 20-Nov-2008
  Multi-center study
  1. Department of Paediatrics, Kashyap Nursing Home, Mumbai.
  2. Department of Paediatrics, KEM Hospital, Pune
  3. Department of Paediatrics, J.K.Lon, SMS Hospital, Jaipur
  4. Panchsheel Hospital, Delhi
Pre-assignment Details: Open-label, single-arm study. Healthy infants between the ages of 6 weeks through exactly 12 weeks (≥42 to ≤84 days) at entry who did not have clinical evidence of active gastrointestinal illness; who did not have fever, with a rectal temperature of greater than and equal to 38 degrees Celsius at first vaccination were enrolled in the study.
Groups:
- RotaTeq™ Vaccine (V260): Subjects enrolled in the study received three doses of RotaTeq™ orally at 3 separate visits 4 to 10 weeks apart.
Period: Overall Study
Arm/Group | RotaTeq™ Vaccine (V260)
Started | 110
Completed | 102
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: Days] | 59.01 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 63
Height [Mean (Standard Deviation); unit: Centimeters] | 57.61 (5.04)
Temperature [Mean (Standard Deviation); unit: Fahrenheit] | 98.58 (0.70)
Weight [Mean (Standard Deviation); unit: Kilograms] | 4.73 (0.71)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Who Exhibit a 3 Fold Rise or Greater From Baseline to Approximately 6 Months in Rotavirus Specific Serum in IgA
Time Frame: Baseline and Approximately 6 Months
Population: The number of subjects contributing to the Full analysis set (FAS) analysis includes all subjects who had immunogenicity data
Measure: Number; unit: Percentage of Participants
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 102
Percentage of Participants | 82.35 [74.95 to 89.75]

2. Primary Outcome: The Percentage of Participants Who Exhibit a 3 Fold Rise or Greater From Baseline to Approximately 6 Months in Rotavirus Specific Serum in IgA
Time Frame: Baseline and Approximately 6 Months
Population: The number of subjects contributing to the per protocol analysis includes all subjects who are not general protocol violators, received all 3 vaccinations at 3 separate visits scheduled at least 4 weeks (28 days) apart and had valid serology results.
Measure: Number; unit: Percentage of Participants
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 99
Percentage of Participants | 82.83 [75.40 to 90.26]

3. Primary Outcome: The Percentage of Participants Who Exihibit 3 Fold Rise Responses or Greater From Baseline to Approximately 6 Months in G1 Serum Neutralizing Antibodies (SNA)
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 102
Percentage of Participants | 38.24 [28.81 to 47.67]

4. Primary Outcome: The Percentage of Participants Who Exihibit 3 Fold Rise Responses or Greater From Baseline to Approximately 6 Months in G2 Serum Neutralizing Antibodies(SNA)
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 102
Percentage of Participants | 14.71 [7.84 to 21.58]

5. Primary Outcome: The Percentage of Participants Who Exihibit 3 Fold Rise Responses or Greater From Baseline to Approximately 6 Months in G3 Serum Neutralizing Antibodies(SNA)
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 102
Percentage of Participants | 30.39 [21.46 to 39.32]

6. Primary Outcome: The Percentage of Participants Who Exihibit 3 Fold Rise Responses or Greater From Baseline to Approximately 6 Months in G4 Serum Neutralizing Antibodies(SNA)
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 102
Percentage of Participants | 37.25 [27.87 to 46.63]

7. Primary Outcome: The Percentage of Participants Who Exihibit 3 Fold Rise Responses or Greater From Baseline to Approximately 6 Months in P1 Serum Neutralizing Antibodies(SNA)
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 102
Percentage of Participants | 30.39 [21.46 to 39.32]

8. Primary Outcome: The Percentage of Participants Who Exihibit 3 Fold Rise Responses or Greater From Baseline to Approximately 6 Months in G1 Serum Neutralizing Antibodies(SNA)
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 99
Percentage of Participants | 37.37 [27.84 to 46.90]

9. Primary Outcome: The Percentage of Participants Who Exihibit 3 Fold Rise Responses or Greater From Baseline to Approximately 6 Months in G2 Serum Neutralizing Antibodies(SNA)
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 99
Percentage of Participants | 14.14 [7.28 to 21.00]

10. Primary Outcome: The Percentage of Participants Who Exihibit 3 Fold Rise Responses or Greater From Baseline to Approximately 6 Months in G3 Serum Neutralizing Antibodies(SNA)
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 99
Percentage of Participants | 29.29 [20.33 to 38.25]

11. Primary Outcome: The Percentage of Participants Who Exihibit 3 Fold Rise Responses or Greater From Baseline to Approximately 6 Months in G4 Serum Neutralizing Antibodies(SNA)
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 99
Percentage of Participants | 35.35 [25.93 to 44.77]

12. Primary Outcome: The Percentage of Participants Who Exihibit 3 Fold Rise Responses or Greater From Baseline to Approximately 6 Months in P1 Serum Neutralizing Antibodies(SNA)
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 99
Percentage of Participants | 29.29 [20.33 to 38.25]

13. Primary Outcome: The Summary of Geometric Mean Titer (GMT) at Baseline & Approximately 6 Months for IgA
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 102
Titer
  IgA GMT at Baseline | 3.81 [2.74 to 5.29]
  IgA GMT at 6 Months | 79.95 [55.23 to 115.73]

14. Primary Outcome: The Summary of Geometric Mean Titer (GMT) at Baseline & Approximately 6 Months for IgA
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 99
Titer
  IgA GMT at Baseline | 3.68 [2.66 to 5.09]
  IgA GMT at 6 Months | 75.12 [51.67 to 109.22]

15. Primary Outcome: The Summary of Geometric Mean Titer (GMT) at Baseline & Approximately 6 Months for G1
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 102
Titer
  G1 GMT at Baseline | 43.53 [35.59 to 53.24]
  G1 GMT at 6 Months | 85.79 [68.65 to 107.20]

16. Primary Outcome: The Summary of Geometric Mean Titer (GMT) at Baseline & Approximately 6 Months for G2
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 102
Titer
  G2 GMT at Baseline | 63.25 [53.46 to 74.83]
  G2 GMT at 6 Months | 50.33 [41.66 to 60.81]

17. Primary Outcome: The Summary of Geometric Mean Titer (GMT) at Baseline & Approximately 6 Months for G3
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 102
Titer
  G3 GMT at Baseline | 27.22 [21.23 to 34.90]
  G3 GMT at 6 Months | 34.32 [26.71 to 44.09]

18. Primary Outcome: The Summary of Geometric Mean Titer (GMT) at Baseline & Approximately 6 Months for G4
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 102
Titer
  G4 GMT at Baseline | 51.91 [43.29 to 62.23]
  G4 GMT at 6 Months | 84.43 [69.36 to 102.79]

19. Primary Outcome: The Summary of Geometric Mean Titer (GMT) at Baseline & Approximately 6 Months for P1
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 102
Titer
  P1 GMT at Baseline | 86.61 [69.48 to 107.95]
  P1 GMT at 6 Months | 104.56 [82.86 to 131.94]

20. Primary Outcome: The Summary of Geometric Mean Titer (GMT) at Baseline & Approximately 6 Months for G1
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 99
Titer
  G1 GMT at Baseline | 43.11 [35.07 to 52.98]
  G1 GMT at 6 Months | 81.19 [65.15 to 101.19]

21. Primary Outcome: The Summary of Geometric Mean Titer (GMT) at Baseline & Approximately 6 Months for G2
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 99
Titer
  G2 GMT at Baseline | 62.91 [52.91 to 74.79]
  G2 GMT at 6 Months | 49.21 [40.62 to 59.61]

22. Primary Outcome: The Summary of Geometric Mean Titer (GMT) at Baseline & Approximately 6 Months for G3
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 99
Titer
  G3 GMT at Baseline | 27.71 [21.48 to 35.73]
  G3 GMT at 6 Months | 32.95 [25.60 to 42.42]

23. Primary Outcome: The Summary of Geometric Mean Titer (GMT) at Baseline & Approximately 6 Months for G4
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 99
Titer
  G4 GMT at Baseline | 51.74 [42.94 to 62.35]
  G4 GMT at 6 Months | 80.88 [65.52 to 98.34]

24. Primary Outcome: The Summary of Geometric Mean Titer (GMT) at Baseline & Approximately 6 Months for P1
Time Frame: Baseline and Approximately 6 Months
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RotaTeq™ Vaccine (V260)
Number analyzed (Participants) | 99
Titer
  P1 GMT at Baseline | 84.17 [67.27 to 105.31]
  P1 GMT at 6 Months | 100.01 [79.28 to 126.15]

ADVERSE EVENTS:
Time Frame: 1. Any SAE/NSAE reported day 1 through day 14 of vaccination 2. Any serious vaccine related AE that occurred throughout the study 3. Any death 4. Any event of clinical interest (intussusception) that occurred throughout the study
Description: Parents/guardians were asked to record AEs on a standardized Vaccine Report Card (VRC) from Day 1 through Day 14 after each dose of RotaTeq™
  Temperatures and any episodes of vomiting and diarrhea were recorded on the card daily from Day 1 through Day 7 after each dose
  6 subjects did not report after dose 1 and were considered lost to follow-up
Arm/Group | RotaTeq™ Vaccine (V260)
Serious Adverse Events (participants affected / at risk) | 1/104
Other Adverse Events (participants affected / at risk) | 47/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq™ Vaccine (V260) (N=104)
Meningitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RotaTeq™ Vaccine (V260) (N=104)
Ear Pain (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 22 (30)
Vomiting (Gastrointestinal disorders) | 19 (29)
Irritability (General disorders) | 1 (2)
Pyrexia (General disorders) | 14 (19)
Meningitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.